CLINICAL TRIAL: NCT04704947
Title: Clinical Study Evaluating Selective or Nonselective Beta Blockers Use and Fracture Risk in Patients With Primary Osteoporosis
Brief Title: Clinical Study Evaluating Beta Blockers Use and Fracture Risk in Patients With Primary Osteoporosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: osteoprosis
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Beta Blocker Toxicity
MeSH Terms: interventions — Propranolol; Bisoprolol; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nonselective beta blocker group (Experimental): Twenty patients with osteoporosis and hypertension on the same treatment as control group in addition to propranolol (Inderal®) 10 mg once daily titrated as patient's response.
  Interventions: Drug: nonselective beta blocker; Drug: alendronate sodium
- cardio-selective beta blocker group (Experimental): Twenty patients with osteoporosis and hypertension on the same treatment as control group in addition to bisoprolol (Concor®) 5 mg once daily titrated as patient's response.
  Interventions: Drug: cardio-selective beta blocker group; Drug: alendronate sodium
- Control group (Placebo Comparator): Ten patient with osteoporosis on alendronate sodium 70 mg (Fosamax®) once/week, vitamin D3 1 mcg once daily and calcium supplement 500 mg once daily.
  Interventions: Drug: alendronate sodium

INTERVENTIONS:
Drug: nonselective beta blocker — nonselective beta blocker
  Other Names: Inderal
  Arms: nonselective beta blocker group
Drug: cardio-selective beta blocker group — cardio-selective beta blocker group
  Other Names: concor
  Arms: cardio-selective beta blocker group
Drug: alendronate sodium — alendronate sodium
  Other Names: alendronate

SUMMARY:
Clinical study evaluating selective or nonselective beta blockers use and fracture risk in patients with primary osteoporosis

DETAILED DESCRIPTION:
Clinical study evaluating selective or nonselective beta blockers use and if there is fracture risk in patients with primary osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* • Male & female osteoporotic patient aged ≥ 50 years

  * Hypertensive & normotensive patients
  * BMD T-score ≥ 2.5 or more SD below peak bone mass

Exclusion Criteria:

* Patients on drugs that may improve osteoporosis disease state such as:

  * Angiotensin converting enzyme inhibitor (ACEI) or Angiotensin receptor blockers (ARBs), Thiazide diuretic, Nitrates, Spironolactone, Statins.

Patients on drugs that may worsen osteoporosis disease state such as:

• Corticosteroids, Loop diuretics, Anticonvulsants, Antidepressants, Aromatase inhibitors, Thyroid replacement therapy and Proton pump inhibitors.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with fracture in each group | 1 year
  the exact number of patients with fracture in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mona Abd El-Rafea Abdo, PH D, Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No